CLINICAL TRIAL: NCT06880692
Title: The Use of Ecological Momentary Assessments to Assess Tick-borne Disease Risk
Brief Title: The Tick App: Changing Behaviors With Educational Messaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of Illinois at Chicago (Other); Michigan State University (Other); Columbia University (Other); Washington State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-0084; 1U01CK000651-01-00 (Other Grant/Funding Number: Centers for Disease Control and Prevention); Protocol Version 9/11/25 (Other: UW Madison); A073600 (Other: UW Madison); 1U01CK000651-01 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Tick Bites
Keywords: tick education; behavior change; tick bite prevention
MeSH Terms: conditions — Tick Bites

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants do not know if they are in the group getting messaging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tick App Educational Materials (Experimental)
  Interventions: Other: Educational Materials delivered via the Tick App
- No Educational Messaging (No Intervention)

INTERVENTIONS:
Other: Educational Materials delivered via the Tick App — Education about tick bite prevention
  Arms: Tick App Educational Materials

SUMMARY:
The goal of this work is to evaluate the use of ecological momentary assessments as a tool to assess risk and risk factors for tick encounters and tick-borne diseases. This study will be conducted across the United States, with a focus the upper Midwest and Northeast and with a focus on Wisconsin and will enroll up to 1000 people.

DETAILED DESCRIPTION:
In the United States, several online and smart-phone apps are available to ID a tick (TickID app, North Carolina State University), submit a picture of a tick (TickSpotters.org, an outreach tool within the larger TickEncounter resource center by the University of Rhode Island) or submit a tick for testing (among other public health agencies, TickReport.com by the University of Massachusetts Amherst). Although these tools are accessible throughout the U.S., they focus on the Northeast. In addition, they do not assess human behavior and tick encounters nor do these tools evaluate prevention and education strategies. A recent study in the Netherlands evaluated the use and effectiveness of a preventative and educational tick app ("Tekenbeet"). This app was well-appreciated, well-used, and improved the user's intention to implement preventative measures. This also illustrates the move of information acquisition from in-hand leaflets to information provision through smartphones.

In this study, data on human behavior regarding tick encounters and tick prevention measures will be obtained from a smartphone application using momentary assessments methodology to assess real time behavior and movement. Ecological momentary assessments are a methodological tool for gathering quantitative behavioral data in real-time, or within the framework of a participant's daily routine.

The daily logs feature provides researchers information about what the participant's activity, location, tick encounters, and prevention measures used. This study will analyze participants who complete 7 daily logs. Their daily logs will be analyzed against the types of educational messaging presented to them within the Tick App.

During a portion of the year the opening screen will contain a prevention message and daily log reminder instead of the home screen. The screen will provide a tick check reminder, a link to the daily log and for half the users the screen will also include a reminder about another prevention behavior (for example bathing/showering). Users will be randomly assigned to the two groups to assess if the additional prevention message increases prevention behavior (tick checks and showering/bathing) and the number of tick encounters.

ELIGIBILITY:
Inclusion Criteria:

* Will to participate in 7 days worth of daily activity logs within the Tick App.
* be able and willing to provide informed consent

Exclusion Criteria:

* Completes less than 7 days worth of daily logs or completes 7+ daily logs but not within 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2020-03-31 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in number of tick prevention behaviors | up to 12 months
  A goal of the intervention is to see an increase in tick prevention behaviors (tick checks and showering). To measure this, the change in number of tick prevention behaviors will be compared between groups. Data collected when participant completes 7 daily logs in app within 12 months.

SECONDARY OUTCOMES:
Change in number of self-reported tick encounters | up to 12 months
  A goal of the intervention is to see a decrease in self-reported tick encounters. To measure this, the change in number of self-reported tick encounters will be compared between groups. Data collected when participant completes 7 daily logs in app within 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Paskewitz, Principal Investigator — University of Wisconsin, Madison; Lyric Bartholomay, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - University of Illinois, Urbana, Illinois
  - Michigan State University, East Lansing, Michigan
  - Columbia University, New York, New York
  - Washington State University, Pullman, Washington

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data collected during the trial, after the deidentification will be available to researchers for independent verification of study outcome or to conduct subsequent clinical research, whose proposed use of the data has been approved by an independent review committee identified for this purpose.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Beginning 9 months after publication of primary outcomes and ending 2 years after that date.
Access Criteria: Proposals should be directed to Susan Paskewitz, smpaskew@wisc.edu or Maria Diuk Wasser, mad2256@columbia.edu. If approved after review by regulatory counsel, requestors will enter into a formal data sharing agreement. Data will be shared via encrypted single-user file transmission protocol.

REFERENCES:
- See also: The Tick App — https://tickapp.us/